CLINICAL TRIAL: NCT06330831
Title: Measuring the Effectiveness of Intensive Group Based CIMT for Young Children
Brief Title: Intensive Group Based CIMT for Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockhurst University (Other)
Collaborators: Ability KC (Unknown)
Responsible Party: Principal Investigator, Katie Ryan-Bloomer, Associate Professor of Occupational Therapy, Rockhurst University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: x2ghr8pc
Record Dates: First submitted 2024-03-05; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hemiplegic Cerebral Palsy; Non-Accidental Traumatic Head Injury to Child
Keywords: Constraint Induced Movement Therapy; Pediatrics; Group Based; Intensive; Young children

STUDY DESIGN:
Intervention Model Description: Study 1 is a single group pre-post study of children who received 1 episode of the intensive, group based CIMT intervention (2 data points- pre CIMT 1 and post CIMT1). Study 2 is a repeated measures design to evaluate the long-term effects of the first episode and the effects of the second episode of intensive group based CIMT (4 data points- pre CIMT1; post CIMT1 (at the end of 1 month intervention); pre CIMT 2- 11 months after post of CIMT1; post CIMT 2- 12 months post CIMT 1)
Masking Description: No masking occurred for the participants or care providers since all parents/caregivers consented to have their children participate in the intensive group based CIMT intervention. The parents/ care providers knew who the interventionists were. The principal investigator was aware of all participants' assignment to the study. The principal investigator also delivered the intervention to the 2-3-year-old group and also served as the assessor of outcomes along with trained student investigators. The principal investigator attempted to limit bias by having all students achieve an inter-rater reliability level of 90% or above (intra-class correlation coefficient ICC>.90) on the QUEST and by not allowing the student investigators or herself to consult the pre-intervention assessment outcome scores until after post-intervention outcome assessment scoring was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive, Group Based CIMT (Experimental): The intensive, group based CIMT program lasted for 3 hours/day x 5 days/week x 4 weeks. Children wore a cast on their non-affected arm for 24 hours/day for 3 weeks. During the last week, the cast was removed to focus on bimanual skills. Occupational therapists ran and were present for every hour of the program. Both physical therapy and speech language pathology cotreated for 1 1/2 hours two times per week and either music, art, or adaptive martial arts occurred 1 hour per week. Interns and volunteers served as intervention assistants to maintain a 2:1 or 1:1 child to therapist/interventionist ratio. The same theme-based lesson plans were used for the 2-3-year-old program and the 4-6-year-old program. Each age group program offered spots for 3-6 children to attend per year except for 2020 when the programs were suspended due to COVID 19 pandemic.
  Interventions: Other: Intensive, Group Based Constraint Induced Therapy (CIMT)

INTERVENTIONS:
Other: Intensive, Group Based Constraint Induced Therapy (CIMT) — See arm description. Children who were in study 2 received two consecutive episodes of the intensive, group based CIMT intervention (episode 1 during the first summer, episode 2 during the following summer).

SUMMARY:
This project aims to investigate the effectiveness of an intensive, group-based Constraint Induced Movement Therapy (CIMT) program for young children ages 2-6 years with unilateral hemiparesis, or weakness on one side of the body. This project involves two studies. Study 1 investigates the effect of one dosage of a 1-month, intensive group based CIMT summer program. Study 2 investigates the effect of a repeated, consecutive episode of the intensive, group based CIMT program for children who attended the program the following summer.

DETAILED DESCRIPTION:
Children with hemiparesis, or weakness on one side of the body, caused by neurological conditions such as cerebral palsy or brain injury often experience difficulty using their arm and hand on their affected side (unilateral function), using both arms together (bimanual coordination) and participating in meaningful activities (occupational performance). Constraint Induced Movement Therapy (CIMT) has become one of the most evidence-based treatments for children with unilateral hemiplegia. Constraint Induced Movement Therapy involves constraining the non-affected arm and hand using a cast or sling to promote the use of the affected hand. Though CIMT offered on an individual basis to children in their own homes has been found to be effective, there are disadvantages to individual, signature models or caregiver delivered models of CIMT which include cost, decreased in number of children who can receive the therapy, and caregiver burden. Group based CIMT offers an alternative model of delivery for CIMT intervention that alleviates some of the challenges. The goal of this overall project was to evaluate the effectiveness of an intensive, group-based Constraint Induced Movement Therapy (CIMT) program for young children ages 20 months through 6 years of age with hemiparesis. The children attended a month-long intensive, group based CIMT program lasting 3 hours/day x 5 days/week x 4 weeks. For the first 3 weeks the children wore a cast on their non-affected arm for nearly 24 hours a day. During the last week of the program, the occupational therapists removed the cast and focused on bimanual skills (using both hands together). The children participated in testing that measured unilateral function (performance of the weaker arm such as range of motion, grasp, ability to bear weight or catch self), bimanual coordination (the ability to use both hands for functional tasks such as holding a toy, cutting food), and occupational performance (the ability to participate in meaningful daily activities- dressing, play, school-related activities). Study 1 analyzed the effects of a single dosage of the CIMT intervention (attending the program for one month). The investigators hypothesized (predicted) that following the study, the children would statistically significantly improve unimanual function, bimanual coordination, and occupational performance. Study 2 analyzed the effects of two, consecutive episodes of CIMT intervention (attending the CIMT program for 2 summers in a row). The researcher hypothesized children would display statistically significant improvements in unimanual function, bimanual coordination, and occupational performance after each episode.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral hemiparesis
* Between the ages of 20 mos.- 6 yrs 11 mos. 30 days
* Authorized through insurance or scholarship to attend the CIMT summer program
* Manual Ability Classification Scale or Mini-MACS level of 1-4
* Able to follow simple commands.

Exclusion Criteria:

* If in child protective service custody since videographic information for QUEST and AHA assessments could not be obtained
* If receiving additional OT therapy during the intensive, group based CIMT program
* If missed more than 3 days of the group based CIMT intervention

Ages: 20 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Quality Upper Extremity Skills Evaluation Test (QUEST) | Study 1: Pre-intervention assessment= within 1 month of start of program, post-intervention = at the end of 1 month program. Study 2: CIMT 2 pre-assessment= 11 months following episode 1 , CIMT 2 post-assessment = 12 months following episode 1
  The Quality Upper Extremity Skills Evaluation Test (QUEST) is a standardized assessment that has the child perform various movements to assess the function of the non-affected arm and the hemiparetic arm in four subtests: Dissociated Movements, Grasps, Weight Bearing and Protective Extension. The children perform reaching, turning forearm over, grasping and releasing of various toys, leaning through their arms in various positions, and catching themselves when tipped out of their base of support in various positions. The QUEST has been standardized with children with unilateral cerebral palsy. Children were videotaped while participating in the QUEST and the principal investigator, clinical investigators, and trained OT students scored the QUEST for this study.
Assisting Hand Assessment (AHA) | Study 1: Pre-intervention assessment= within 1 month of start of program, post-intervention = at the end of 1 month program. Study 2: CIMT 2 pre-assessment= 11 months following episode 1 , CIMT 2 post-assessment = 12 months following episode 1
  The Assisting Hand Assessment (AHA) is a standardized criterion test which measures children's ability to use the affected hand as an assisting hand when manipulating numerous toys that require two hands. The AHA is a play-based assessment where the children video recorded while playing with various toys. A certified AHA rater (which the principal investigator is) reviews the video and scores the children on 22 items. A total sum score and scaled score percentile can be generated. The AHA Kids version was standardized on children 18 months to 12 years of age on children with cerebral palsy and brachioplexus injury. The AHA has been used in numerous research studies and shows good responsiveness to change in performance from before to after intervention.
Canadian Occupational Performance Measure (COPM) | Study 1: Pre-intervention assessment= within 1 month of start of program, post-intervention = at the end of 1 month program. Study 2: CIMT 2 pre-assessment= 11 months following episode 1 , CIMT 2 post-assessment = 12 months following episode 1
  The Canadian Occupational Performance Measure (COPM) is a standardized assessment that measures occupational performance of and satisfaction of performance of meaningful, individualized goals. Clients identify five most important areas of occupational difficulty within the domains of self-care, productivity, and leisure. Parents of children under the age of 8 years, rate the child's performance on a scale of one (poor performance) to 10 (nearly perfect performance) and satisfaction of one (not satisfied at all) to 10 (very satisfied). The scores for performance and satisfaction can be summed to give a performance total and satisfaction total. Many studies have demonstrated the COPM displays good responsiveness to change, meaning this assessment can easily detect change in performance and satisfaction from before to after intervention.
Pediatric Evaluation Disability Inventory (PEDI) | Study 1: Pre-intervention assessment= within 1 month of start of program, post-intervention = at the end of 1 month program. Study 2: CIMT 2 pre-assessment= 11 months following episode 1 , CIMT 2 post-assessment = 12 months following episode 1
  The Pediatric Evaluation Disability Inventory (PEDI) assesses children's functional skill ability within the domains of selfcare, mobility, and social function. The parents rate a child's performance as capable or unable on discrete skills within each domain. The parents also rate the level of assistance they provide the child on the Caregiver Assistance Scale from total assistance to none (child independence). The caregivers also rate the level of modifications needed for each subdomain. The original PEDI was standardized on children with and without disabilities from 6 months to 7 1/2 years of age. The PEDI has been used in other CIMT studies as a measure of occupational performance with some responsivity. Only the selfcare and social function domains were used for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S Ryan-Bloomer, Principal Investigator — Associate Professor of OT Rockhurst University; Occupational Therapist at Ability KC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorley M, Lannin N, Cusick A, Novak I, Boyd R. Reliability of the quality of upper extremity skills test for children with cerebral palsy aged 2 to 12 years. Phys Occup Ther Pediatr. 2012 Feb;32(1):4-21. doi: 10.3109/01942638.2011.602389. Epub 2011 Aug 15. PMID 21838618
- [Background] Krumlinde-Sundholm L, Holmefur M, Kottorp A, Eliasson AC. The Assisting Hand Assessment: current evidence of validity, reliability, and responsiveness to change. Dev Med Child Neurol. 2007 Apr;49(4):259-64. doi: 10.1111/j.1469-8749.2007.00259.x. PMID 17376135
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] McColl MA, Denis CB, Douglas KL, Gilmour J, Haveman N, Petersen M, Presswell B, Law M. A Clinically Significant Difference on the COPM: A Review. Can J Occup Ther. 2023 Mar;90(1):92-102. doi: 10.1177/00084174221142177. Epub 2023 Jan 17. PMID 36650928
- [Background] James S, Ziviani J, Boyd R. A systematic review of activities of daily living measures for children and adolescents with cerebral palsy. Dev Med Child Neurol. 2014 Mar;56(3):233-44. doi: 10.1111/dmcn.12226. Epub 2013 Aug 13. PMID 23937056
- [Background] Regalado A, Decker B, Flaherty BM, Zimmer L, Brown I. Effectiveness of Constraint-Induced Movement Therapy for Children With Hemiparesis Associated With Cerebral Palsy: A Systematic Review. Am J Occup Ther. 2023 May 1;77(3):7703205160. doi: 10.5014/ajot.2023.050152. PMID 37358836
- [Background] Chiu HC, Ada L. Constraint-induced movement therapy improves upper limb activity and participation in hemiplegic cerebral palsy: a systematic review. J Physiother. 2016 Jul;62(3):130-7. doi: 10.1016/j.jphys.2016.05.013. Epub 2016 Jun 17. PMID 27323932
- [Background] Tinderholt Myrhaug H, Ostensjo S, Larun L, Odgaard-Jensen J, Jahnsen R. Intensive training of motor function and functional skills among young children with cerebral palsy: a systematic review and meta-analysis. BMC Pediatr. 2014 Dec 5;14:292. doi: 10.1186/s12887-014-0292-5. PMID 25475608
- [Background] Walker C, Shierk A, Roberts H. Constraint Induced Movement Therapy in Infants and Toddlers with Hemiplegic Cerebral Palsy: A Scoping Review. Occup Ther Health Care. 2022 Jan;36(1):29-45. doi: 10.1080/07380577.2021.1953206. Epub 2021 Aug 2. PMID 34339315
- [Background] Wang TN, Liang KJ, Liu YC, Shieh JY, Chen HL. Effects of Intensive Versus Distributed Constraint-Induced Movement Therapy for Children With Unilateral Cerebral Palsy: A Quasi-Randomized Trial. Neurorehabil Neural Repair. 2023 Feb-Mar;37(2-3):109-118. doi: 10.1177/15459683231162330. Epub 2023 Mar 28. PMID 36987387
- [Background] Wu WC, Hung JW, Tseng CY, Huang YC. Group constraint-induced movement therapy for children with hemiplegic cerebral palsy: a pilot study. Am J Occup Ther. 2013 Mar-Apr;67(2):201-8. doi: 10.5014/ajot.2013.004374. PMID 23433275
- [Background] Gelkop N, Burshtein DG, Lahav A, Brezner A, Al-Oraibi S, Ferre CL, Gordon AM. Efficacy of constraint-induced movement therapy and bimanual training in children with hemiplegic cerebral palsy in an educational setting. Phys Occup Ther Pediatr. 2015 Feb;35(1):24-39. doi: 10.3109/01942638.2014.925027. Epub 2014 Jul 1. PMID 24983295
- [Background] Cohen-Holzer M, Katz-Leurer M, Reinstein R, Rotem H, Meyer S. The effect of combining daily restraint with bimanual intensive therapy in children with hemiparetic cerebral palsy: a self-control study. NeuroRehabilitation. 2011;29(1):29-36. doi: 10.3233/NRE-2011-0674. PMID 21876293